CLINICAL TRIAL: NCT00760799
Title: Randomized Study of Anular Repair With the Xclose Tissue Repair System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anulex Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06101_B
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Diskectomy
Keywords: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Diskectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard discectomy without anular repair
  Interventions: Procedure: Discectomy with anular repair
- 2 (Experimental): Standard Discectomy with anular repair
  Interventions: Procedure: Discectomy with anular repair

INTERVENTIONS:
Procedure: Discectomy with anular repair — Comparison of discectomy with and without repair to the anulus fibrosus of the intervertebral disc
  Other Names: Repair of the anulus fibrosus following discectomy.

SUMMARY:
The purpose of this study is to evaluate the benefits of anulus fibrosus repair utilizing Xclose™ compared to a discectomy without anulus fibrosus repair.

DETAILED DESCRIPTION:
Discectomy surgery is intended to remove the impinging fragment on the nerve root thus alleviating the pain and providing the nerve with a better healing environment. Discectomy procedures entail removing a bony portion of the vertebral body to access the posterior side of the disc space, and then removing the impinging fragment from the disc. The fragment being removed can either be contained within the wall of the anulus, which requires incision into the anulus to remove it, or it could be extruded through an anular fissure. In the absence of a safe and easy method to close or seal the defect in the anulus following a discectomy procedure, surgeons are left with no alternative but to leave the anulus in this compromised state which is largely the current practice. This rent in the soft tissue of the anulus fibrosus can lead to postoperative problems if the remaining nuclear tissue in the disc pushes through the anular defect or incision causing recurrent or persistent pain.

Initial studies involved the placement of sutures to seal the anular defect. This work strongly suggested that microsurgical anular reconstruction can reduce recurrent herniations and re-operations, post discectomy. Unfortunately, this technique is not easy to perform and may pose an increased risk to the patient.

This study utilizes the Xclose™ Tissue Repair System to re-approximate the compromised tissue of the anulus fibrosus in appropriately randomized patients in an effort to quantify the benefits of anular repair for discectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for a one or two level discectomy
* Positive imaging evidence of intervertebral disc herniation at location corresponding to patient's radicular signs or symptoms
* Anular tear or slit incision and additionally deemed to include sufficient tissue for tissue reapproximation
* Persistent and predominant radicular pain
* Pre-operative leg pain score > 4.0 cm on a 10 cm Visual Analog Scale (VAS)
* Leg pain unresponsive to conservative treatment (physical therapy and non-steroidal anti-inflammatory medical therapy) for 6 or more weeks; exception, individuals suffering from acute and uncontrollable severe leg pain
* Patient is willing and able to comply with study requirements; willing and able to sign a study-specific, informed consent form, complete necessary study paperwork and return for required follow-up visits.

Exclusion Criteria:

* Age less than 18 years
* Prior or planned surgical procedure intended to fuse or stabilize the lumbar spine
* Previous surgery involving index level
* Cauda Equina Syndrome
* Evidence of severe disc degeneration
* Greater than Grade I spondylolisthesis or retrolisthesis at the affected level
* No apparent anular defect and no indication to open the anulus at time of procedure
* Active local or systemic infection
* Active malignancy or other significant medical co-morbidities
* Current chemical dependency or significant emotional and/or psychosocial disturbance that would impact treatment outcome or study participation
* Patient or legal guardians who are unwilling or unable to cooperate or give written informed consent
* Women who are pregnant or with child bearing potential and who are not on a reliable form of birth control
* Current fracture, tumor and/or deformity (> 15° of lumbar scoliosis, using Cobb measuring technique) of the spine
* Documented history of allergy or intolerance to PET
* Patient is currently enrolled in other research that could confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2007-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Re-operations due to re-herniation (repeat discectomy procedure) | 2 wks and at 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Patient outcomes (utilizing Oswestry Disability Index, Visual Analog Scale and SF-12 quality of life assessment), Health care utilization, Return to work | 2 weeks and at 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - North Alabama Neurological, P.A., Huntsville, Alabama
  - Texas Back Institute, Phoenix, Arizona
  - Desert Institute for Spine Care, Phoenix, Arizona
  - University of California San Diego, San Diego, California
  - Denver Spine (Porter Hospital), Greenwood Village, Colorado
  - Denver Spine (Presbyterian/St. Luke's Hospital), Greenwood Village, Colorado
  - North Florida Regional Hospital, Gainesville, Florida
  - Lyerly Neurosurgical (Baptist Health), Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Lyerly Neurosurgical (Centerone), Jacksonville, Florida
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Chicago Institute of Neurosurgery and Neuroresearch, Chicago, Illinois
  - Palos Community Hospital, Palos Heights, Illinois
  - Indiana Spine Group, Indianapolis, Indiana
  - Heartland Spine, Overland Park, Kansas
  - New England Baptist, Boston, Massachusetts
  - Oakwood Hospital, Dearborn, Michigan
  - Henry Ford, Detroit, Michigan
  - Central Minnesota Neurosciences, Sartell, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hudson Valley Neurosurgical Associates, Suffern, New York
  - Capital Neurosurgery, Raleigh, North Carolina
  - Atlantic Neurosurgical & Spine, Wilmington, North Carolina
  - Pennsylvania Spine Institute, Harrisburg, Pennsylvania
  - West Penn Neurosurgery Group, Pittsburgh, Pennsylvania
  - Our Lady of Fatima Hospital, North Providence, Rhode Island
  - East Tennessee Brain and Spine, Johnson City, Tennessee
  - Texas Back Institute, Plano, Texas
  - San Antonio Orthopedic Group, San Antonio, Texas
  - South Texas Spine Clinic, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wyoming Spine and Neurosurgery Associates, Cheyenne, Wyoming

REFERENCES:
- [Derived] Bailey A, Araghi A, Blumenthal S, Huffmon GV; Anular Repair Clinical Study Group. Prospective, multicenter, randomized, controlled study of anular repair in lumbar discectomy: two-year follow-up. Spine (Phila Pa 1976). 2013 Jun 15;38(14):1161-9. doi: 10.1097/BRS.0b013e31828b2e2f. PMID 23392414